CLINICAL TRIAL: NCT06060015
Title: Effect of Subarachnoid Hyperbaric Bupivacaine on Mean Arterial Pressure in Obese Pregnant Patients Undergoing Cesarean Section
Brief Title: Effect of Subarachnoid Hyperbaric Bupivacaine in Obese Pregnant Patients Undergoing Cesarean Section
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, María de los Angeles Campechano Ascencio, Anestesiologist, Hospital Civil de Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 168/23
Record Dates: First submitted 2023-09-08; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Anesthesia; Obstetric Anesthesia Problems
Keywords: Anesthesia; Obesity; Cesarean; Subarachnoid; Bupivacaine; pregnancy
MeSH Terms: conditions — Obesity | interventions — Bupivacaine; Glucose

STUDY DESIGN:
Intervention Model Description: Clinical trial open controlled parallel randomized simple
Who Masked: Participant, Investigator
Masking Description: You do not know the dose of bupivacaine you receive
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5mg bupivacaine (Experimental): Anesthetic technique, the patient receives subarachnoid hyperbaric bupivacaine at a dose of 5mg
  Interventions: Drug: 5mg bupivacaine
- 10mg bupivacaine (Experimental): Anesthetic technique, the patient receives subarachnoid hyperbaric bupivacaine at a dose of 10mg
  Interventions: Drug: 10mg bupivacaine

INTERVENTIONS:
Drug: 5mg bupivacaine — Anesthetic technique, the patient receives subarachnoid hyperbaric bupivacaine at a dose of 5mg
  Other Names: hyperbaric bupivacaine 1ml; bupivacaine/Dextrose 1ml
  Arms: 5mg bupivacaine
Drug: 10mg bupivacaine — Anesthetic technique, the patient receives subarachnoid hyperbaric bupivacaine at a dose of 10 mg
  Other Names: hyperbaric bupivacaine 2ml; bupivacaine/Dextrose 2ml
  Arms: 10mg bupivacaine

SUMMARY:
Evaluates the effect of hyperbaric subarachnoid bupivacaine at doses of 5 mg vs 10 mg on mean arterial pressure in obese pregnant patients undergoing cesarean section

DETAILED DESCRIPTION:
Patients over 18 years of age, with a pregnancy of ≥37 weeks of gestation and adequate fetal well-being, with obesity with a BMI ≥30 kg/m2 presented for cesarean surgery will be included in the study. The objectives of the study protocol, benefits, and benefits will be explained to them. and risks and by election by sealed envelope will be assigned to one of the two study groups, they will be given to sign the consent letter under information. They underwent pre-anesthetic evaluation, baseline vital signs: non-invasive blood pressure, mean arterial pressure (MAP), O2 saturation and heart rate, fetal heart rate will be recorded from the fetal monitor. A preload of Hartmann's solution fluids at 10ml/kg of pre-pregnancy weight and premedication with omeprazole 40mg and metoclopramide 10mg will be administered. Once inside the operating room, baseline vital signs will be recorded and the placement of anesthesia with mixed technique neuraxial block (epidural catheter placement + subarachnoid block) will begin in a sitting position, the anatomical reference of the intervertebral space L2-L3, L3- will be located. L4. The aseptic and antiseptic technique with povidone-iodine and alcohol will be performed on the skin, sterile fields will be placed, the skin and subcutaneous tissue will be infiltrated with 5 ml of 2% lidocaine, a Tuohy No. 17 needle is inserted with the "hanging Drop" technique, to locate the epidural space, it was corroborated with the "loss of resistance" technique. Through the "Tuohy needle", the "spinal needle" No. 27 spinal needle is inserted until cerebrospinal fluid (CSF) is obtained. The blocking dose of hyperbaric bupivacaine of 10 mg (2 ml) or mg (1 ml) will be administered according to the assigned group; The "spinal needle" was withdrawn and the epidural catheter was inserted in a cephalic direction, leaving 5 cm inside the epidural space. The catheter was fixed to the skin with adhesive tape for later use. The patient will be placed in the supine position and a position is given with the surgical table 30 degrees to the left. Vital sign monitoring was started every 3 minutes for the first 15 minutes and then every 5 minutes until the end of the procedure. When a MAP record of less than 20% is obtained at the beginning, 10 mg ephedrine will be administered, an evaluation of the sensory block will begin 6 minutes after administering the block dose, with the prick technique, this evaluation will be It will be performed every 3 minutes during the first 15 minutes and then every 15 minutes until the end of the surgery. Simultaneously, an assessment of motor blockade will begin with a Bromage scale. After taking the second vital signs (3 minutes), the patient will be asked if she feels nauseated or if she vomits and it will be recorded. At the time of the extraction of the fetus, the Apgar score given by the neonatologist at one minute and at 5 minutes of extrauterine life will be recorded. Once the placenta has been delivered, a sample for gasometry will be taken with a heparinized syringe from the umbilical artery and sent to the laboratory for processing. A dose of local anesthetic will be administered through a 5% to 2% lidocaine epidural catheter if the patient reports discomfort or pain and the surgical procedure has not been completed. The information collected will be recorded in the data collection sheet. The sample size was calculated with a formula for comparing two means with a finite population.A pilot test was carried out with the specified criteria, which included 40 patients, 20 patients received 5 mg of subarachnoid hyperbaric bupivacaine and 20 patients received 10 mg, for the maximum arterial hypotension variable registered a standard deviation of 16.87 was obtained. The finite population was obtained by registering the total cesarean sections of the Civil Hospital of Guadalajara performed during the year 2022, which were 1,256 cesarean sections and losses of 20% are calculated, obtaining a total of 53 patients per group with a total of 106 patients. Once the sample is completed, the database will be started in the Microsoft Office Excel program, which will be exported to the statistical program Statistics Product and Service Solution (SPSS) for statistical analysis. The data obtained will be expressed through measures of central tendency and dispersion, mean, minimum, maximum, median and standard deviation for quantitative variables, and frequencies and percentages in the case of qualitative variables. The intragroup differences for the quantitative variables were performed using the Student's T test, differences between the groups were determined with the U Mann Whitney test. Qualitative variables will be analyzed with the Chi Square test. A value of p≤0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy ≥37 weeks gestation with single fetus
* Body mass index (BMI) ≥ 30 kg/m2
* Indication of termination of pregnancy via abdominal caesarean section
* Indication of subarachnoid neuraxial block under mixed technique
* Signing of consent under information

Exclusion Criteria:

* Allergy to local anesthetics
* Psychiatric treatment (antidepressants, anxiolytics, antipsychotics)
* Addiction to any type of drug
* Liver, renal, pulmonary or cardiac disease
* High blood pressure
* Type I, II and gestational diabetes
* Diagnostic of non-calming fetal state

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Single fetus and pregnancy whit BMI≥ 30 kg/m2
Enrollment: 106 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Assess the mean blood pressure | 3 hour
  Number of pregnant patients with obesity who present a decrease in mean arterial pressure after the administration of subarachnoid hyperbaric bupivacaine with doses of 5mg and 10mg during cesarean surgery
Determine the effects on the heart rate | 3 hour
  Number of pregnant patients with obesity who present changes in heart rate such as bradycardia (heart rate less than 60 beats minute) or tachycardia (heart rate greater than 120 beats minute) after administration of subarachnoid hyperbaric bupivacaine with doses of 5mg and 10 mg during cesarean surgery
Determine the effects on the O2 saturation | 3 hour
  Number of pregnant patients with obesity who present changes in O2 saturation after administration of subarachnoid hyperbaric bupivacaine with doses of 5mg and 10mg during cesarean surgery

SECONDARY OUTCOMES:
Describe the adverse effects (nausea or vomiting) | 3 hour
  Number of pregnant patients with obesity with side effects such as nausea or vomiting after administration of subarachnoid hyperbaric bupivacaine with doses of 5mg and 10 mg during cesarean surgery
Identify the level of sensory blockade | 15 minutes
  Number of pregnant patients with obesity with adequate sensory block (thoracic dermatome 4 is defined as adequate to begin the surgical technique), the level of sensory block reached after the administration of subarachnoid hyperbaric bupivacaine with doses of 5mg and 10mg. The sensory block was evaluated using pinprick. Every 3 minutes the first 15 minutes after the subarachnoid block.
Describe the adverse effects on the fetus | 1 hour
  Number of pregnant patients with obesity with any side effect associated with the fetal bradycardia anesthetic technique (Fetal heart rate less than 120 beats minute) cardiac arrest (Fetal heart rate less than 100 beats minute) And in the newborn fetal acidosis (umbilical vein gasometry with Hydrogen Potential (pH) <7.0 or excess bases >-12 mmol/L)
Document the Apgar score | 5 minutes
  Document the Apgar score in the newborn. (Apgar Score evaluate five sign: color, heart rate, reflex irritability, muscle tone and respiration) The score ranges from 0 to 2 per sign according to the criteria of the neonatologist, to grant a maximum score of 10 points. A grade of less than 7 points is considered low Apgar scores. This scores is registered t minute and five minutes of life.

CONTACTS AND LOCATIONS:
Overall Officials: María de los Angeles Campechano Ascencio, MSc, Principal Investigator — Hospital Civil de Guadalajara; Miriam Mendez del Villar, PhD, Study Director — Universidad de Guadalajara Centro Universitario de Tonalá; Leonel Garcia Benavides, PhD, Study Chair — Universidad de Guadalajara Centro Universitario de Tonalá; Jorge Bravo Rubio, MSc, Study Chair — Hospital Civil de Guadalajara; Edy David Rubio Arellano, MSc, Study Chair — Universidad de Guadalajara Centro Universitario Ciencias de la Salud
Locations (1):
- Hospital Civil de Guadalajara, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eltzschig HK, Lieberman ES, Camann WR. Regional anesthesia and analgesia for labor and delivery. N Engl J Med. 2003 Jan 23;348(4):319-32. doi: 10.1056/NEJMra021276. No abstract available. PMID 12540646
- [Result] Badve MH, Golfeiz C, Vallejo MC. Anesthetic considerations for the morbid obese parturient. Int Anesthesiol Clin. 2014 Summer;52(3):132-47. doi: 10.1097/AIA.0000000000000024. No abstract available. PMID 24946047
- [Result] Tonidandel A, Booth J, D'Angelo R, Harris L, Tonidandel S. Anesthetic and obstetric outcomes in morbidly obese parturients: a 20-year follow-up retrospective cohort study. Int J Obstet Anesth. 2014 Nov;23(4):357-64. doi: 10.1016/j.ijoa.2014.05.004. Epub 2014 Jun 4. PMID 25201313
- [Result] Ouzounian JG, Elkayam U. Physiologic changes during normal pregnancy and delivery. Cardiol Clin. 2012 Aug;30(3):317-29. doi: 10.1016/j.ccl.2012.05.004. Epub 2012 Jun 20. PMID 22813360
- [Result] Hood DD, Dewan DM. Anesthetic and obstetric outcome in morbidly obese parturients. Anesthesiology. 1993 Dec;79(6):1210-8. doi: 10.1097/00000542-199312000-00011. PMID 8267196
- [Result] Tan T, Sia AT. Anesthesia considerations in the obese gravida. Semin Perinatol. 2011 Dec;35(6):350-5. doi: 10.1053/j.semperi.2011.05.021. PMID 22108086
- [Result] Ngan Kee WD, Khaw KS, Tan PE, Ng FF, Karmakar MK. Placental transfer and fetal metabolic effects of phenylephrine and ephedrine during spinal anesthesia for cesarean delivery. Anesthesiology. 2009 Sep;111(3):506-12. doi: 10.1097/ALN.0b013e3181b160a3. PMID 19672175
- [Result] Lee Y, Balki M, Parkes R, Carvalho JC. Dose requirement of intrathecal bupivacaine for cesarean delivery is similar in obese and normal weight women. Rev Bras Anestesiol. 2009 Nov-Dec;59(6):674-83. doi: 10.1016/s0034-7094(09)70092-3. English, Portuguese. PMID 20011857
- [Result] Carvalho B, Collins J, Drover DR, Atkinson Ralls L, Riley ET. ED(50) and ED(95) of intrathecal bupivacaine in morbidly obese patients undergoing cesarean delivery. Anesthesiology. 2011 Mar;114(3):529-35. doi: 10.1097/ALN.0b013e318209a92d. PMID 21307769
- [Result] Reyes M, Pan PH. Very low-dose spinal anesthesia for cesarean section in a morbidly obese preeclamptic patient and its potential implications. Int J Obstet Anesth. 2004 Apr;13(2):99-102. doi: 10.1016/j.ijoa.2003.09.004. PMID 15321413
- [Result] Teoh WH, Thomas E, Tan HM. Ultra-low dose combined spinal-epidural anesthesia with intrathecal bupivacaine 3.75 mg for cesarean delivery: a randomized controlled trial. Int J Obstet Anesth. 2006 Oct;15(4):273-8. doi: 10.1016/j.ijoa.2006.03.004. Epub 2006 Jun 13. PMID 16774830
- [Result] Bamgbade OA, Khalaf WM, Ajai O, Sharma R, Chidambaram V, Madhavan G. Obstetric anaesthesia outcome in obese and non-obese parturients undergoing caesarean delivery: an observational study. Int J Obstet Anesth. 2009 Jul;18(3):221-5. doi: 10.1016/j.ijoa.2008.07.013. Epub 2009 May 17. PMID 19447599
- [Result] Nani FS, Torres ML. Correlation between the body mass index (BMI) of pregnant women and the development of hypotension after spinal anesthesia for cesarean section. Rev Bras Anestesiol. 2011 Jan-Feb;61(1):21-30. doi: 10.1016/S0034-7094(11)70003-4. PMID 21334504
- [Result] Ngaka TC, Coetzee JF, Dyer RA. The Influence of Body Mass Index on Sensorimotor Block and Vasopressor Requirement During Spinal Anesthesia for Elective Cesarean Delivery. Anesth Analg. 2016 Dec;123(6):1527-1534. doi: 10.1213/ANE.0000000000001568. PMID 27870737
- [Result] Hassanin AS, El-Shahawy HF, Hussain SH, Bahaa Eldin AM, Elhawary MM, Elbakery M, Elsafty MSE. Impact of interval between induction of spinal anesthesia to delivery on umbilical arterial cord ph of neonates delivered by elective cesarean section. BMC Pregnancy Childbirth. 2022 Mar 17;22(1):216. doi: 10.1186/s12884-022-04536-y. PMID 35300620
- [Result] Klohr S, Roth R, Hofmann T, Rossaint R, Heesen M. Definitions of hypotension after spinal anaesthesia for caesarean section: literature search and application to parturients. Acta Anaesthesiol Scand. 2010 Sep;54(8):909-21. doi: 10.1111/j.1399-6576.2010.02239.x. Epub 2010 Apr 23. PMID 20455872
- [Result] Zhu T, Tang J, Zhao F, Qu Y, Mu D. Association between maternal obesity and offspring Apgar score or cord pH: a systematic review and meta-analysis. Sci Rep. 2015 Dec 22;5:18386. doi: 10.1038/srep18386. PMID 26692415
- [Result] Soens MA, Birnbach DJ, Ranasinghe JS, van Zundert A. Obstetric anesthesia for the obese and morbidly obese patient: an ounce of prevention is worth more than a pound of treatment. Acta Anaesthesiol Scand. 2008 Jan;52(1):6-19. doi: 10.1111/j.1399-6576.2007.01483.x. PMID 18173431
- [Result] Ring LE. The anesthetic approach to operative delivery of the extremely obese parturient. Semin Perinatol. 2014 Oct;38(6):341-8. doi: 10.1053/j.semperi.2014.07.008. Epub 2014 Aug 19. PMID 25146109
- [Result] Kominiarek MA, Chauhan SP. Obesity Before, During, and After Pregnancy: A Review and Comparison of Five National Guidelines. Am J Perinatol. 2016 Apr;33(5):433-41. doi: 10.1055/s-0035-1567856. Epub 2015 Nov 20. PMID 26588260
- [Result] Silva JC, Amaral AR, Ferreira BD, Petry JF, Silva MR, Krelling PC. [Obesity during pregnancy: gestational complications and birth outcomes.]. Rev Bras Ginecol Obstet. 2014 Nov;36(11):509-513. doi: 10.1590/s0100-720320140005024. Epub 2014 Nov 1. Portuguese. PMID 25493403
- [Result] Lamon AM, Habib AS. Managing anesthesia for cesarean section in obese patients: current perspectives. Local Reg Anesth. 2016 Aug 16;9:45-57. doi: 10.2147/LRA.S64279. eCollection 2016. PMID 27574464
- [Result] Dennis AT, Castro JM, Ong M, Carr C. Haemodynamics in obese pregnant women. Int J Obstet Anesth. 2012 Apr;21(2):129-34. doi: 10.1016/j.ijoa.2011.11.007. Epub 2012 Feb 11. PMID 22326199
- [Result] Rodrigues FR, Brandao MJ. Regional anesthesia for cesarean section in obese pregnant women: a retrospective study. Rev Bras Anestesiol. 2011 Jan-Feb;61(1):13-20. doi: 10.1016/S0034-7094(11)70002-2. PMID 21334503
- [Result] Wise RA, Polito AJ, Krishnan V. Respiratory physiologic changes in pregnancy. Immunol Allergy Clin North Am. 2006 Feb;26(1):1-12. doi: 10.1016/j.iac.2005.10.004. PMID 16443140
- [Result] Kim ST. Anesthetic management of obese and morbidly obese parturients. Anesth Pain Med (Seoul). 2021 Oct;16(4):313-321. doi: 10.17085/apm.21090. Epub 2021 Oct 29. PMID 35139612
- [Result] Chandra S, Tripathi AK, Mishra S, Amzarul M, Vaish AK. Physiological changes in hematological parameters during pregnancy. Indian J Hematol Blood Transfus. 2012 Sep;28(3):144-6. doi: 10.1007/s12288-012-0175-6. Epub 2012 Jul 15. PMID 23997449
- [Result] American College of Obstetricians and Gynecologists. ACOG Committee opinion no. 549: obesity in pregnancy. Obstet Gynecol. 2013 Jan;121(1):213-7. doi: 10.1097/01.aog.0000425667.10377.60. PMID 23262963
- [Result] Gaiser R. Anesthetic Considerations in the Obese Parturient. Clin Obstet Gynecol. 2016 Mar;59(1):193-203. doi: 10.1097/GRF.0000000000000180. PMID 26694495
- [Result] Arias J, Lacassie HJ. [Prophylaxis and treatment of arterial hypotension during caesarean with spinal anaesthesia]. Rev Esp Anestesiol Reanim. 2013 Nov;60(9):511-8. doi: 10.1016/j.redar.2012.07.023. Epub 2012 Oct 23. Spanish. PMID 23092743
- [Result] Davies GAL, Maxwell C, McLeod L. No. 239-Obesity in Pregnancy. J Obstet Gynaecol Can. 2018 Aug;40(8):e630-e639. doi: 10.1016/j.jogc.2018.05.018. PMID 30103887
- [Result] Rasolonjatovo TY, Ravololonirina BM, Randriamanantany ZA, Raveloson NE. [Spinal anesthesia for cesarean section: risk factors for emergence of Apgar scores below 7 in Malagasy newborns]. Pan Afr Med J. 2014 Oct 23;19:193. doi: 10.11604/pamj.2014.19.193.3392. eCollection 2014. French. PMID 25821536
- [Result] Mercier FJ, Auge M, Hoffmann C, Fischer C, Le Gouez A. Maternal hypotension during spinal anesthesia for caesarean delivery. Minerva Anestesiol. 2013 Jan;79(1):62-73. Epub 2012 Nov 18. PMID 23135692
- [Result] Polin CM, Hale B, Mauritz AA, Habib AS, Jones CA, Strouch ZY, Dominguez JE. Anesthetic management of super-morbidly obese parturients for cesarean delivery with a double neuraxial catheter technique: a case series. Int J Obstet Anesth. 2015 Aug;24(3):276-80. doi: 10.1016/j.ijoa.2015.04.001. Epub 2015 Apr 8. PMID 25936783
- [Result] Sng BL, Siddiqui FJ, Leong WL, Assam PN, Chan ES, Tan KH, Sia AT. Hyperbaric versus isobaric bupivacaine for spinal anaesthesia for caesarean section. Cochrane Database Syst Rev. 2016 Sep 15;9(9):CD005143. doi: 10.1002/14651858.CD005143.pub3. PMID 27629425
- [Result] Lamon AM, Einhorn LM, Cooter M, Habib AS. The impact of body mass index on the risk of high spinal block in parturients undergoing cesarean delivery: a retrospective cohort study. J Anesth. 2017 Aug;31(4):552-558. doi: 10.1007/s00540-017-2352-0. Epub 2017 Apr 18. PMID 28421314
- [Result] Edwards RK, Cantu J, Cliver S, Biggio JR Jr, Owen J, Tita ATN. The association of maternal obesity with fetal pH and base deficit at cesarean delivery. Obstet Gynecol. 2013 Aug;122(2 Pt 1):262-267. doi: 10.1097/AOG.0b013e31829b1e62. PMID 23969793
- [Result] Hollowell J, Pillas D, Rowe R, Linsell L, Knight M, Brocklehurst P. The impact of maternal obesity on intrapartum outcomes in otherwise low risk women: secondary analysis of the Birthplace national prospective cohort study. BJOG. 2014 Feb;121(3):343-55. doi: 10.1111/1471-0528.12437. Epub 2013 Sep 11. PMID 24034832
- [Result] Committee Membership:; Burns S, Biering-Sorensen F, Donovan W, Graves DE, Jha A, Johansen M, Jones L, Krassioukov A, Kirshblum S, Mulcahey MJ, Read MS, Waring W. International standards for neurological classification of spinal cord injury, revised 2011. Top Spinal Cord Inj Rehabil. 2012 Winter;18(1):85-99. doi: 10.1310/sci1801-85. No abstract available. PMID 23460761
- See also: World Health Organization. Obesity and Overweight Descriptive note No 311. — http://www.who.int/mediacentre/factsheets/fs311/es/